CLINICAL TRIAL: NCT00396461
Title: Phase IV-IV. ICULIP,a Prospective,Multi-centre,Randomised,Comparative,Double-blind Study to Evaluate Two Different Types of Lipid Emulsions Used for Total Parenteral Nutrition in Critical Patients and Their Influence on Nosocomial Infection.
Brief Title: ICULIP, Influence of Two Lipid Emulsions in the Nosocomial Infection in Critical Patients
Acronym: ICULIP
Status: Terminated | Phase: Phase 4 | Type: Interventional
Sponsor: B. Braun Medical SA (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HC-G-H-0510; 2005-003542-33 (EudraCT Number)
Record Dates: First submitted 2006-11-03; First posted 2006-11-07 (Estimated); Last update posted 2013-07-19 (Estimated); Status verified 2013-07

CONDITIONS: Critical Illness
Keywords: Critical Illness; Fat Emulsions, Intravenous; Superinfection; Parenteral Nutrition
MeSH Terms: conditions — Critical Illness; Superinfection; Hyperphagia

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- TPN A (Group I) (Active Comparator): Emulsion based on 20% MCT/LCT (50:50 ratio)
  Interventions: Drug: MCT/LCT (1:1)
- TPN B (Group II) (Experimental): Emulsion based on 20% MCT/LCT/w3 (50:40:10 ratio), medium- and long-chain triglycerides and fish oil triglycerides
  Interventions: Drug: MCT/LCT/omega-3 (5:4:1)

INTERVENTIONS:
Drug: MCT/LCT (1:1) — Emulsion based on 20% MCT/LCT (50:50 ratio)
  Other Names: LIPOFUNDINA
  Arms: TPN A (Group I)
Drug: MCT/LCT/omega-3 (5:4:1) — Emulsion based on 20% MCT/LCT/w3 (50:40:10 ratio), medium- and long-chain triglycerides and fish oil triglycerides.
  Other Names: LIPOPLUS
  Arms: TPN B (Group II)

SUMMARY:
This study aims to analyse the effect of two total parenteral nutrition diets with lipid emulsions of different compositions on the incidence of nosocomial infection in critical patients. One diet will contain an MCT/LCT emulsion concentrated to 20% (50:50 ratio) and the other will comprise an MCT/LCT/fish oil emulsion (50:40:10 ratio). The secondary objective of this study is to analyse mortality in hospital and up to 6 months of discharge.

DETAILED DESCRIPTION:
During the last years the most widely used lipid emulsion for parenteral nutrition has been based on soybean oil. This first generation of lipid emulsions used in TPN contained w-6 series polyunsaturated long-chain fatty acids (LCT) from soy, maize, sunflower and safflower oil. LCT contain an excess of linoleic acid which, when metabolised, produce large quantities of arachidonic acid and its metabolites. Although the generally used doses seem safe (1-2 g/kg/day by continuous perfusion), alterations in pulmonary function in patients with acute adult respiratory distress syndrome have been described, as have alterations in platelet function, hepatic function and haemodynamics, which are attributed to the excess of said metabolites. However, the most important side effect of the LCT lipid infusions is its influence on the immune response. Experimental and clinical studies show that LCT can interfere with various stages of the immune response such as the production of antibodies, complement synthesis, granulocytic and lymphocytic activity and the reticuloendothelial system. Various hypotheses have been formulated to explain the modulator effect of the polyunsaturated fatty acids on immune function: changes in the permeability of the cellular membrane, modifications in the synthesis of eicosanoids and the presence of peroxides derived from the oxidation of polyunsaturated fatty acids.

In summary, although linoleic acid as a dietary essential fatty acid is important, its excessive intake is associated with undesirable immunological and inflammatory events. Thus it is recommended that soybean oil should be partly replaced by other lipids.

To avoid these side effects the second generation lipid emulsions were developed. These contain a combination of medium- and long-chain fatty acids (MCT/LCT) with lower w-6 fatty acid content. MCT/LCT lipid emulsions are safe and do not produce biochemical or metabolic alterations or gaseous exchange in patients with ARDS. MCT/LCT combinations seem to reduce the generation of eicosanoids and do not alter the immune response in in-vitro and experimental studies. The impact of these differences on the nosocomial infection and the clinical prognosis of the patients has not been studied sufficiently despite the fact that some studies show reduced mortality and morbidity using MCT/LCT emulsions when compared with the use of pure LCT emulsions. MCT/LCT emulsions are normally used in clinical practice on patients that have required parenteral nutrition for 20 years.

Recently, the clinical use in artificial nutrition of omega-3 series polyunsaturated fatty acids, eicosapentaenoic acid (EPA) and docosahexaenoic acid (DHA) present in many fish oils has been significant. EPA is a precursor to certain eicosanoid series that compensate the proinflammatory effects of the eicosanoids in arachidonic acid (omega-6 series). The objective is immunomodulation to attenuate the inflammatory response of patients without negatively impacting on the immune function. The use of enteral diets enriched with omega-3 series fatty acids (fish oil) in post-operation cancer patients showed a reduction in the number of days in hospital and infectious complications.

The use of fish oil or fat emulsions enriched with fish oil (omega-3) in parenteral nutrition has already been the subject of various studies: where modulation of the inflammatory response markers has been shown, reduces the stay in hospital and the need for mechanical ventilation in patients undergoing major abdominal surgery, reduces the stay in hospital in patients undergoing digestive surgery… So, w-3 lipids exhibit strong immunologic properties. They offer the possibility to counterbalance the negative effects of conventional w-6 fatty acids. Recent studies exhibit positive effects of intravenous use of fish oil on immunologic functions and clinical parameters in surgical and septic patients

The purpose of this study is to analyse the effect of two total parenteral nutrition diets with lipid emulsions of different compositions on the incidence of nosocomial infection in critical patients. One diet will contain an MCT/LCT emulsion concentrated to 20% (50:50 ratio) (w3:w6 is 1:7) and the other will comprise an MCT/LCT/fish oil emulsion (50:40:10 ratio) (w3:w6 is 1:2,7). The secondary objective of this study is to analyse mortality in hospital and up to 6 months after discharge.

ELIGIBILITY:
INCLUSION CRITERIA:

Patients of both sexes, prospective admission to Intensive Care Units (ICUs), over 18 years, where TPN is required as a nutritional metabolic support for a minimum period of 5 days and where said patients have signed the informed consent form.

The indications for administration of parenteral nutrition shall be those recommended by the American Society of Parenteral and Enteral Nutrition (ASPEN), and in particular:

* Severe malnutrition
* Major intra-abdominal surgery
* Peritonitis
* Intestinal ischaemia
* Intestinal occlusion
* Gastrointestinal fistulas
* Small intestine

Patients of both sexes, over 18 years, that commencing nutritional support with enteral diets in the first 3 days of admission to ICU require parenteral nutrition as:

* 75% of the calculated energy requirements have not been reached after three days receiving enteral nutrition.
* Gastrointestinal complications have been suffered as a result of enteral nutrition that cannot be treated or are persistent in the first 3 days of admission.

In this case EN will be suspended and the patient will be included in the protocol receiving PN.

EXCLUSION CRITERIA:

* APACHE II < 13
* Morbid obesity (BMI ≥ 39)
* Hepatic disease defined within the following set of parameters:

  1. Portal hypertension with gastrointestinal bleeding on admission
  2. Clinically apparent hepatocellular ascites
  3. Hepatocellular bilirubin higher than 3 mg/dL
  4. Serum albumin less than 30 g/L with portal hypertension
  5. Grade II or higher encephalopathy
  6. Clinical diagnosis of alcoholic hepatitis
* Chronic renal insufficiency defined by one of the following criteria:

  1. Plasmatic creatinine greater than 4 mg/dL
  2. Chronic peritoneal dialysis or haemodialysis
* Patients with severe acquired or familial hyperlipidaemias (> 400 mg/day) of any kind
* Serious chronic neurological disease defined by one of the following criteria:

  1. Cerebrovascular accident with persistent neurological deficit in the past six months
  2. Neurological deficit that necessitates chronic confinement
* Neoplastic patients with metastasis and a life expectancy of less than six months
* Patients that underwent chemotherapy or radiotherapy during the month prior to the study
* Patients that received chronic treatment with corticoids in the month preceding admission to ICU. Patients receiving treatment with corticoids since admission to ICU for septic shock should not be excluded.
* Continuous infusion treatment for more than 24 hours with propofol or with other pharmaceuticals where lipid emulsions are used as the vehicle
* Infectious diseases transmitted through the blood, products derived from blood or urine: hepatitis B, C and HIV
* Inclusion in another clinical trial
* Having received TPN in the month prior to inclusion in the study
* Pregnancy
* Refusal to participate in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 212 (Estimated)
Dates: Start 2006-11; Primary Completion 2010-09 (Actual); Study Completion 2011-02 (Actual)

PRIMARY OUTCOMES:
The analyses will particularly focus on: Pneumonia associated with mechanical ventilation, Catheter infection, Bacteraemia not associated with catheter, Urinary infection, Infection of surgical wounds and Intra-abdominal abscess and peritonitis. | Patients will receive at least 5 days of PN. Clinical condition and nosocomial infection will be monitored daily until the first phase of the study is completed on day 28 or the patient is discharged from the unit.
Compare the incidence of nosocomial infection associated with the administration of two different lipid solutions in total parenteral nutrition of patients in an Intensive Care Unit. | Patients will receive at least 5 days of PN. Clinical condition and nosocomial infection will be monitored daily until the first phase of the study is completed on day 28 or the patient is discharged from the unit.

SECONDARY OUTCOMES:
Study mortality at the end of the study and 6 months after discharge from ICU; Hospital stay and/or in Intensive Care Unit; Mechanical ventilation days; Assessment of hepatic function; Assessment of nutritional efficacy. | At the end of the study and 6 months after discharge from ICU.

CONTACTS AND LOCATIONS:
Overall Officials: Abelardo García de Lorenzo, MD, Study Chair — Hospital Universitario La Paz; Alfonso Bonet Saris, MD_Study Coordinator, Principal Investigator — University Hospital of Girona Dr. Josep Trueta; Teodoro Grau Carmona, MD_Study Coordinator, Study Chair — Hospital Severo Ochoa Leganés (Madrid)
Locations (22):
- Spain (22):
  - Hospital General Universitario de Alicante, Alicante, Alicante
  - Hospital Son Dureta, Palma de Mallorca, Balearic Islands
  - Hospital del Mar (Institut Municipal d'Assistència Sanitària, IMAS), Barcelona, Barcelona
  - Hospital Universitari Vall d'Hebrón, Barcelona, Barcelona
  - Hospital Universitario de Bellvitge (H.U.B.), L'Hospitalet de Llobregat, Barcelona
  - Hospital de Cruces, Barakaldo, Bizcaya
  - Hospital Universitario Marqués de Valdecilla, Santander, Cantabria
  - Hospital Universitario "Puerta del Mar", Cadiz, Cádiz
  - Hospital Universitari de Girona Doctor Josep Trueta, Girona, Girona
  - Hospital Universitario de Gran Canaria Dr. Negrín, Las Palmas de Gran Canaria, Gran Canaria
  - Complejo Hospitalario Materno Insular de Gran Canaria, Las Palmas de Gran Canaria, Gran Canaria
  - Hospital Universitario Virgen de las Nieves, Granada, Granada
  - Hospital Universitario Arnau de Vilanova, Lleida, Lleida
  - Hospital Severo Ochoa, Leganés, Madrid
  - Fundación Jiménez Díaz, Madrid, Madrid
  - Hospital Universitario "Virgen de la Arrixaca", El Palmar, Murcia
  - Hospital General Universitario "Reina Sofía", Murcia, Murcia
  - Hospital Regional Universitario Carlos Haya, Málaga, Málaga
  - Hospital Universitario de Valme, Seville, Sevilla
  - Hospital Clínico Universitario de Valencia, Valencia, Valencia
  - Hospital Universitario Del Río Hortega, Valladolid, Valladolid
  - Hospital Universitario Miguel Servet, Zaragoza, Zaragoza

REFERENCES:
- [Background] Cerra FB. Hypermetabolism, organ failure, and metabolic support. Surgery. 1987 Jan;101(1):1-14. PMID 3541266
- [Background] Garcia-de-Lorenzo A. Lipid emulsions with different phospholipid/triglyceride ratio in critically ill septic and traumatic patients. Crit Care Med. 1998 Dec;26(12):2094-5. doi: 10.1097/00003246-199812000-00049. No abstract available. PMID 9875927
- [Background] Bach AC, Frey A, Lutz O. Clinical and experimental effects of medium-chain-triglyceride-based fat emulsions--a review. Clin Nutr. 1989 Oct;8(5):223-35. doi: 10.1016/0261-5614(89)90032-0. PMID 16837294
- [Background] Mathru M, Dries DJ, Zecca A, Fareed J, Rooney MW, Rao TL. Effect of fast vs slow intralipid infusion on gas exchange, pulmonary hemodynamics, and prostaglandin metabolism. Chest. 1991 Feb;99(2):426-9. doi: 10.1378/chest.99.2.426. PMID 1989806
- [Background] Gogos CA, Kalfarentzos F. Total parenteral nutrition and immune system activity: a review. Nutrition. 1995 Jul-Aug;11(4):339-44. PMID 8580573
- [Background] Calder PC, Sherrington EJ, Askanazi J, Newsholme EA. Inhibition of lymphocyte proliferation in vitro by two lipid emulsions with different fatty acid compositions. Clin Nutr. 1994 Apr;13(2):69-74. doi: 10.1016/0261-5614(94)90062-0. PMID 16843362
- [Background] Clarke PJ, Ball MJ, Hands LJ, Dennison AR, Tunbridge A, White K, Kettlewell MG. Use of a lipid containing medium chain triglycerides in patients receiving TPN: a randomized prospective trial. Br J Surg. 1987 Aug;74(8):701-4. doi: 10.1002/bjs.1800740818. PMID 3115354
- [Background] Barton RG. Nutrition support in critical illness. Nutr Clin Pract. 1994 Aug;9(4):127-39. doi: 10.1177/0115426594009004127. PMID 8078451
- [Background] Suchner U, Katz DP, Furst P, Beck K, Felbinger TW, Senftleben U, Thiel M, Goetz AE, Peter K. Effects of intravenous fat emulsions on lung function in patients with acute respiratory distress syndrome or sepsis. Crit Care Med. 2001 Aug;29(8):1569-74. doi: 10.1097/00003246-200108000-00012. PMID 11505129
- [Background] Gogos CA, Kalfarentzos FE, Zoumbos NC. Effect of different types of total parenteral nutrition on T-lymphocyte subpopulations and NK cells. Am J Clin Nutr. 1990 Jan;51(1):119-22. doi: 10.1093/ajcn/51.1.119. PMID 2136970
- [Background] Jensen GL, Mascioli EA, Seidner DL, Istfan NW, Domnitch AM, Selleck K, Babayan VK, Blackburn GL, Bistrian BR. Parenteral infusion of long- and medium-chain triglycerides and reticuloendothelial system function in man. JPEN J Parenter Enteral Nutr. 1990 Sep-Oct;14(5):467-71. doi: 10.1177/0148607190014005467. PMID 2122019
- [Background] Suchner U, Senftleben U. Immune modulation by polyunsaturated fatty acids during nutritional therapy: interactions with synthesis and effects of eicosanoids. Infusionsther Transfusionsmed. 1994 Jun;21(3):167-82. doi: 10.1159/000222968. PMID 7919904
- [Background] Calder PC. Long-chain n-3 fatty acids and inflammation: potential application in surgical and trauma patients. Braz J Med Biol Res. 2003 Apr;36(4):433-46. doi: 10.1590/s0100-879x2003000400004. Epub 2003 Apr 8. PMID 12700820
- [Background] Gadek JE, DeMichele SJ, Karlstad MD, Pacht ER, Donahoe M, Albertson TE, Van Hoozen C, Wennberg AK, Nelson JL, Noursalehi M. Effect of enteral feeding with eicosapentaenoic acid, gamma-linolenic acid, and antioxidants in patients with acute respiratory distress syndrome. Enteral Nutrition in ARDS Study Group. Crit Care Med. 1999 Aug;27(8):1409-20. doi: 10.1097/00003246-199908000-00001. PMID 10470743
- [Background] Weiss G, Meyer F, Matthies B, Pross M, Koenig W, Lippert H. Immunomodulation by perioperative administration of n-3 fatty acids. Br J Nutr. 2002 Jan;87 Suppl 1:S89-94. doi: 10.1079/bjn2001461. PMID 11895158
- [Background] Koller M, Senkal M, Kemen M, Konig W, Zumtobel V, Muhr G. Impact of omega-3 fatty acid enriched TPN on leukotriene synthesis by leukocytes after major surgery. Clin Nutr. 2003 Feb;22(1):59-64. doi: 10.1054/clnu.2002.0592. PMID 12553951
- [Background] Tsekos E, Reuter C, Stehle P, Boeden G. Perioperative administration of parenteral fish oil supplements in a routine clinical setting improves patient outcome after major abdominal surgery. Clin Nutr. 2004 Jun;23(3):325-30. doi: 10.1016/j.clnu.2003.07.008. PMID 15158295
- [Background] ASPEN Board of Directors: Guidelines for the use of parenteral and enteral nutrition in adults and pediatric patients. JPEN 2001
- [Background] Carpentier YA, Van Gossum A, Dubois D, Deckeibaum R. Lipid Metabolism in Parenteral Nutrition. In: Wilmore DW, Carpentier YA (Eds). Metabolic Support of the Critically III Patient. Berlin, Springer-Veriag 1993, pp 35-74
- [Background] Driscoll DF, Adolph M, Bistrian BR. Lipid emulsions in parenteral nutrition. In: Rombeau JL, Rolandelli R, eds. Parenteral nutrition. Philadelphia: W. B. Saunders Company; 2000:35-39.
- [Background] Santoli D, Zurier RB. Prostaglandin E precursor fatty acids inhibit human IL-2 production by a prostaglandin E-independent mechanism. J Immunol. 1989 Aug 15;143(4):1303-9. PMID 2545787
- [Background] Kinsella JE, Lokesh B. Dietary lipids, eicosanoids, and the immune system. Crit Care Med. 1990 Feb;18(2 Suppl):S94-113. No abstract available. PMID 2105185
- [Background] Kumar SG, Das UN, Kumar KV, Madhavi N, Das NP, Tan BKH. Effect of n-6 and n-3 fatty acids on the proliferation of human lymphocyes and their secretion of TN F-alpha and IL-2 in vitro. Nutr Res 1992; 12: 815-823.
- [Background] Grau T, Ruiz de Adana JC, Zubillaga S, Fuerte S, Giron C. [Randomized study of two different fat emulsions in total parenteral nutrition of malnourished surgical patients;effect of infectious morbidity and mortality]. Nutr Hosp. 2003 May-Jun;18(3):159-66. Spanish. PMID 12875092
- [Background] Grimminger F, Seeger W, Mayer K. Use of n-3 fatty acid-containing lipid emulsions in the intensive care unit environment: the clinician's view. Clinical Nutrition 2002, 21, Supplement 2: 23-29.
- [Background] Wichmann MW, Morlion B, Czarnetzki H-D, Thul P, Jauch K-W. Reduction of length of postoperative stay by fish oil containing lipid emulsion - data from a multicenter trial. Clinical Nutrition 2004, 23: 1471
- See also: Spanish Society for Parenteral and Enteral Nutrition — http://www.senpe.com
- See also: ASPEN, American Society for Parenteral and Enteral Nutrition --> Nutrition-related Links — http://www.nutritioncare.org/
- See also: Spanish Society for Intensive Medicine, Critical and Coronary Units — http://www.semicyuc.org/